CLINICAL TRIAL: NCT00601835
Title: Immunogenicity and Safety of Canadian Manufactured Tetanus and Diphtheria Toxoids Adsorbed (Td) for Adult Use Vaccine Compared With U.S. Manufactured Tetanus and Diphtheria Toxoids Adsorbed for Adult Use Vaccine In Persons 60 Years of Age and Older and Immunogenicity and Safety of Canadian Td Vaccine in Persons 11 Through 59 Years of Age
Brief Title: Canadian Manufactured Tetanus and Diphtheria Toxoids Adsorbed (Td) Vaccine Compared With U.S. Manufactured Td
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: TDC01
Record Dates: First submitted 2008-01-15; First posted 2008-01-28 (Estimated); Results first posted 2011-02-18 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Diphtheria; Tetanus
Keywords: Diphtheria; Tetanus
MeSH Terms: conditions — Diphtheria; Tetanus | interventions — Tetanus Toxoid; Vaccines; Diphtheria-Tetanus Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Canadian Td Vaccine Group (Experimental): Participants received Canadian manufactured Td vaccine
  Interventions: Biological: Tetanus and Diphtheria Toxoids Adsorbed (Td) Vaccine
- United States Td Vaccine Group (Active Comparator): Participants received US manufactured Td vaccine
  Interventions: Biological: Tetanus and Diphtheria Toxoids Adsorbed (Td) Vaccine

INTERVENTIONS:
Biological: Tetanus and Diphtheria Toxoids Adsorbed (Td) Vaccine — 0.5 mL, Intramuscular, single dose
  Other Names: TENIVAC™
  Arms: Canadian Td Vaccine Group
Biological: Tetanus and Diphtheria Toxoids Adsorbed (Td) Vaccine — 0.5 mL, Intramuscular, Single dose
  Other Names: DECAVAC®
  Arms: United States Td Vaccine Group

SUMMARY:
To compare the seroprotection rates and booster responses to Canadian-manufactured Tetanus and Diphtheria Toxoids Adsorbed vaccine to the seroprotection rates and booster responses to the US-manufactured Tetanus and Diphtheria Toxoids Adsorbed vaccine when administered to subjects ≥ 60 years of age.

To compare the post-vaccination geometric mean titers of antibody (GMTs) to Canadian manufactured Tetanus and Diphtheria Toxoids Adsorbed vaccine to the post-vaccination GMTs to the US manufactured Tetanus and Diphtheria Toxoids Adsorbed vaccine when administered to subjects ≥ 60 years of age.

DETAILED DESCRIPTION:
This is a multi-center, partially open-label, partially randomized double blind trial for immunogenicity and safety in the United States. Participants will be enrolled to one of three treatment groups:

* Subjects ages 11-59 years will receive Canadian manufactured Td vaccine on Day 0
* Subjects 60 years or older will be randomized to receive either US manufactured Td on Day 0, or,
* Subjects 60 years or older randomized to receive Canadian manufactured Td on Day 0

The trial is designed to assess the safety of Canadian Manufactured Tetanus and Diphtheria Toxoids Adsorbed vaccine in all trial participants 11 to 59 years of age and to describe the immune responses in subsets of adolescents (11-14, and 15-18 years of age) and in a subset of adults 19-59 years of age. The trial will also compare the immune responses and safety in subjects ≥ 60 years of age receiving Canadian Manufactured Tetanus and Diphtheria Toxoids Adsorbed vaccine to an equal number of subjects ≥ 60 years of age receiving US Manufactured Tetanus and Diphtheria Toxoids Adsorbed vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Participant is healthy as per medical history reported by subject.
* Participant is at least 11 years of age at the time of vaccination.
* Participant has a signed Institutional Review Board (IRB)-approved informed assent/consent form. For subjects 11 to 17 years of age, a written informed consent must be obtained from parent(s) or legal guardian(s) and a written informed assent must be obtained from the subject
* Participant provides history or documentation of primary or booster immunization with Diphtheria and Tetanus.
* Female participants of childbearing potential must have a negative urine pregnancy test at the time of enrollment.

Exclusion Criteria:

* Serious and uncontrolled chronic disease (i.e., cardiac, pulmonary, renal, neurologic, metabolic, rheumatologic, etc.).
* Known or suspected impairment of immunologic function.
* Acute medical illness with or without fever within the last 72 hours or an oral temperature ≥ 100.4°F (≥ 38°C) at the time of enrollment.
* Administration of immune globulin or other blood products within the last three months; administration of corticosteroids (injected or oral) or other immunomodulatory therapy within six weeks of the study vaccine. However, individuals on a tapering dose schedule of oral steroids may be included in the trial, as long as steroids were discontinued more than two weeks prior to enrollment.
* Received any vaccine, other than influenza vaccine, in the 28-day period prior to enrollment or scheduled to receive any vaccination, other than influenza prior to Visit 2 blood draw. For influenza vaccine only, exclude if received in the 14 day period prior to enrollment or scheduled to receive in the 14 day period after Visit 1.
* Suspected or known hypersensitivity to Td components, thimerosal (for subjects > 60 years of age) or latex rubber.
* Unable to attend scheduled visits or unable to comply with the study procedures.
* Enrolled in another clinical trial.
* Any condition that would pose a health risk to the participant or interfere with the evaluation of the vaccine in the opinion of the investigator.
* A positive urine pregnancy test at the time of enrollment for all females of childbearing potential.
* Female of childbearing potential who does not agree either to remain abstinent or to use effective birth control during the period of the trial.
* Breast feeding during the period of the trial.
* A history of Guillain- Barré syndrome within 6 weeks after a previous dose of a tetanus toxoid-containing vaccine.
* Receipt of a tetanus or diphtheria vaccination within the 5 years prior to enrollment.
* A previous history of diphtheria disease within the last 25 years or tetanus disease
* History of Arthus-type hypersensitivity reaction or a temperature >103° F following a prior dose of tetanus toxoid, unless 10 years have elapsed since the previous dose.

Ages: 11 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 3651 (Actual)
Dates: Start 2004-05; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (2):
- United States (2):
  - Oakland, California
  - Pittsburgh, Pennsylvania

REFERENCES:
- See also: http://www.sanofipasteur.com — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in the study from 06 May 2004 through 13 December 2004, in 2 medical sites (4 investigators) in the US.
Pre-assignment Details: A total of 3,651 participants that met the inclusion and exclusion criteria were enrolled in the study. One participant declined vaccination.
  The immunogenicity subsets consist of all participants ≥ 60 years of age; the safety subsets consist of all participants ≥ 60 years of age and one third of participants 11 to 59 years of age.
Groups:
- Canadian Td Vaccine Group: Participants received the Canadian manufactured Tetanus and Diphtheria Toxoids Adsorbed vaccine for Adult Use (TENIVAC™)
- United States Td Vaccine Group: Participants received the US manufactured Tetanus and Diphtheria Toxoids Adsorbed vaccine for Adult Use (DECAVAC®)
Period: Overall Study
Arm/Group | Canadian Td Vaccine Group | United States Td Vaccine Group
Started | 2950 | 700
Completed | 2890 | 686
Not Completed | 60 | 14
Not completed — Withdrawal by Subject | 9 | 6
Not completed — Physician Decision | 1 | 0
Not completed — Lost to Follow-up | 37 | 5
Not completed — Adverse Event | 1 | 1
Not completed — Relocate | 12 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Canadian Td Vaccine Group | United States Td Vaccine Group | Total
Number analyzed (Participants) | 2950 | 700 | 3650
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1501 | 0 | 1501
  Between 18 and 65 years | 1000 | 257 | 1257
  >=65 years | 449 | 443 | 892
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.6 (23.49) | 69.3 (7.89) | 40.5 (25.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1629 | 403 | 2032
  Male | 1321 | 297 | 1618
Region of Enrollment [Number; unit: participants]
  United States | 2950 | 700 | 3650

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants ≥ 60 Years of Age With Antibody Levels ≥ 0.10 IU/mL to Tetanus and Diphtheria.
Description: Seroprotection and booster responses for both tetanus and diphtheria were considered to be an antibody level of ≥ 0.10 IU/mL 28 days post-vaccination with either the Canadian-manufactured Tetanus and Diphtheria Toxoids Adsorbed vaccine or the US-manufactured Tetanus and Diphtheria Toxoids Adsorbed vaccine in participants ≥ 60 years of age.
Time Frame: 28 Days post-vaccination
Population: Seroprotection and Booster Responses to Tetanus and Diphtheria were determined in subjects ≥ 60 years of age in the per-protocol immunogenicity population.
Measure: Number; unit: Percentage of participants
Arm/Group | Canadian Td Vaccine Group | United States Td Vaccine Group
Number analyzed (Participants) | 661 | 658
Percentage of participants
  Tetanus Post-vaccination Seroprotection | 96 | 97
  Diphtheria Post-vaccination Seroprotection | 71 | 71
  Tetanus Booster Response | 82 | 84
  Diphtheria Booster Response | 66 | 63

2. Secondary Outcome: Post-vaccination Geometric Mean Titer (GMT) to Tetanus and Diphtheria in Participants ≥ 60 Years Vaccinated With Canadian-manufactured or US-manufactured Tetanus and Diphtheria Toxoids Adsorbed Vaccine.
Time Frame: 28 Days post-vaccination
Population: Geometric mean titers were determined in subjects ≥ 60 years of age in the per-protocol immunogenicity population
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Canadian Td Vaccine Group | United States Td Vaccine Group
Number analyzed (Participants) | 661 | 658
Titers
  Tetanus post-vaccination | 6.83 [6.01 to 7.77] | 7.35 [6.54 to 8.26]
  Diphtheria post-vaccination | 0.459 [0.371 to 0.567] | 0.409 [0.332 to 0.504]

3. Other Pre Specified Outcome: Number of Participants Reporting Solicited Injection Site and Systemic Reactions Post-vaccination With Canadian-Manufactured or US-Manufactured Tetanus and Diphtheria Toxoids Adsorbed Vaccine.
Description: Solicited injection site reactions: Pain, Redness, and Swelling. Solicited systemic reactions: Chills, Diarrhea, Fever (temperature), Headache, Malaise, Muscle weakness, Nausea, Pain in joints, Rash, and Vomiting.
Time Frame: 0-14 days post-vaccination
Population: Solicited safety parameters were in all enrolled and vaccinated participants ≥ 60 years of age and one third of participants 11 to 59 years of age. A subset of the intend-to-treat population.
Measure: Number; unit: Participants
Arm/Group | Canadian Td Vaccine Group | United States Td Vaccine Group
Number analyzed (Participants) | 1450 | 700
Participants
  Any Injection site pain | 832 | 209
  Grade 3 Injection site pain (require medical care) | 7 | 5
  Any Injection site redness | 299 | 132
  Grade 3 Injection site redness (≥ 50 mm) | 28 | 20
  Any Injection site swelling | 205 | 93
  Grade 3 Injection site swelling (≥ 50 mm) | 32 | 11
  Any Chills | 80 | 32
  Grade 3 Chills (Incapacitating) | 5 | 2
  Any Diarrhea | 152 | 53
  Grade 3 Diarrhea (≥ 5 episodes) | 6 | 1
  Any Fever | 95 | 40
  Grade 3 Fever (≥ 39.0 °C) | 2 | 1
  Any Headache | 380 | 122
  Grade 3 Headache (Incapacitating) | 16 | 4
  Any Malaise | 226 | 90
  Grade 3 Malaise (Incapacitating) | 13 | 6
  Any Muscle weakness | 267 | 61
  Grade 3 Muscle weakness (Incapacitating) | 6 | 2
  Any Nausea | 106 | 34
  Grade 3 Nausea (Incapacitating) | 6 | 1
  Any Pain in joints | 201 | 74
  Grade 3 Pain in joints (Incapacitating) | 7 | 1
  Any Vomiting | 33 | 6
  Grade 3 Vomiting (≥ 3 episodes) | 6 | 1

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 6 months post-vaccination in all participants enrolled in the study.
Arm/Group | Canadian Td Vaccine Group | United States Td Vaccine Group
Serious Adverse Events (participants affected / at risk) | 58/2950 | 44/700
Other Adverse Events (participants affected / at risk) | 832/2950 | 209/700
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Canadian Td Vaccine Group (N=2950) | United States Td Vaccine Group (N=700)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2)
Angina pectoris (Cardiac disorders) | 1 (1) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 2 (2)
Moebius II syndrome (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Thyroid mass (Endocrine disorders) | 0 (0) | 1 (1)
Retinal artery occlusion (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Colonic polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal achalasia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peritonitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectocele (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 2 (2) | 4 (4)
Death (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis acute (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 2 (2) | 0 (0)
Gangrene (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Infectious mononucleosis (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hepatic trauma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip Fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Colon Cacer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Paraganglion neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1)
Guillain-Barre syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Post-traumatic headache (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Calculus ureteric (Renal and urinary disorders) | 0 (0) | 1 (1)
Cystocele (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Urethral obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Endometriosis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pelvic prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Chronic obstructive pulmonary disease exacerbated (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive airways disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Arterial rupture (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Canadian Td Vaccine Group (N=2950) | United States Td Vaccine Group (N=700)
Injection site pain (General disorders) | 832/1434 (832) | 209/693 (209)
Injection site redness (General disorders) | 299/1434 (299) | 132/693 (132)
Injection site swelling (General disorders) | 205/1434 (205) | 93/693 (93)
Chills (General disorders) | 80/1434 (80) | 32/693 (32)
Diarrhea (Gastrointestinal disorders) | 152/1434 (152) | 53/693 (53)
Pyrexia (General disorders) | 95/1427 (95) | 40/687 (40)
Headache (Nervous system disorders) | 380/1434 (380) | 122/693 (122)
Malaise (General disorders) | 226/1433 (226) | 90/692 (90)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 267/1434 (267) | 61/692 (61)
Nausea (Gastrointestinal disorders) | 106/1434 (106) | 34/692 (34)
Pains in joints (Musculoskeletal and connective tissue disorders) | 201/1434 (201) | 74/693 (74)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.